CLINICAL TRIAL: NCT00640718
Title: Evaluation of EarlySense EverOn™ System in Medical / Surgical Ward
Brief Title: Evaluation of EverOn™ System in Medical / Surgical Ward
Status: Withdrawn | Type: Observational
Sponsor: EarlySense Ltd. (Industry)
Responsible Party: Dalia Argaman, EarlySense Ltd
Other Study IDs: ES-MRK-PROT1.1
Record Dates: First submitted 2008-03-17; First posted 2008-03-21 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2008-03

CONDITIONS: Post Operative Patient; Patients Requiring PCA; Respiratory Patients; Patients in Risk of Fall
Keywords: heart and respiratory monitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The EverOn™ system developed by EarlySense, Ltd., the sponsor of this study, is intended to assist hospitals to better address and improve recognition and response to changes in a patient's condition.

The system, monitors the patient while in bed consists of a contact-free sensor that is placed under the bed mattress and identifies respiratory and heart rates, degree of patient's movement or agitation while in bed as well as patient's actual exit out of the bed. The EverOn system does not require a physical contact with the patient, eliminating the need for any direct contact electrodes, leads, cuffs or nasal cannulae.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years.
2. Patients not monitored continuously by telemetry, vital sign monitor or oximetry.
3. Patients not requiring special mattresses (e.g. airflow).
4. The patient or a legal guardian is ready to sign the Informed Consent.

Exclusion Criteria:

1. Patients that at the judgment of the staff in the evaluating unit, are not able to communicate coherently and respond to nurses' questions.
2. Patients monitored continuously by telemetry, vital sign monitor or oximetry.
3. Patients requiring special mattresses.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults hospitalized in medical surgical units and are willing to sign consent form
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Estimated); Study Completion 2010-05 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- MetroWest Medical Center, Framingham, Massachusetts, United States

REFERENCES:
- See also: Institute for Health Care Improvement (IHI) — http://www.ihi.org/ihi